CLINICAL TRIAL: NCT00602277
Title: A Phase 1 Study of Reovirus Serotype 3 - Dearing Strain (REOLYSIN®) (NSC 729968) in Patients With Ovarian, Primary Peritoneal and Fallopian Tube Carcinoma
Brief Title: Viral Therapy in Treating Patients With Ovarian Epithelial Cancer, Primary Peritoneal Cancer, or Fallopian Tube Cancer That Did Not Respond to Platinum Chemotherapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00234; NCI-2009-00234 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000584038; OSU-07022; 2007C0028; 07022 (Other: Ohio State University Comprehensive Cancer Center); 7853 (Other: CTEP); P30CA016058 (NIH); U01CA076576 (NIH)
Record Dates: First submitted 2008-01-19; First posted 2008-01-28 (Estimated); Last update posted 2016-08-08 (Estimated); Status verified 2016-08

CONDITIONS: Recurrent Fallopian Tube Carcinoma; Recurrent Ovarian Carcinoma; Recurrent Primary Peritoneal Carcinoma
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — reolysin

ARMS (1):
- Treatment (viral therapy) (Experimental): Patients receive wild-type reovirus IV over 60 minutes on days 1-5 in course 1, followed by insertion of an IP access port. Beginning in course 2, patients receive wild-type reovirus IV over 60 minutes on days 1-5 and wild-type reovirus IP over 10 minutes on days 1 and 2*. Treatment with IV and IP wild-type reovirus repeats every 28 days in the absence of disease progression or unacceptable toxicity. (phase II closed as of 1/7/2011). NOTE: *Patients receive IP wild-type reovirus on days 2 and 3 in course 3.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Wild-type Reovirus

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Wild-type Reovirus
  Other Names: Reolysin

SUMMARY:
This phase I/II trial is studying the side effects and best dose of viral therapy in treating patients with ovarian epithelial cancer, primary peritoneal cancer, or fallopian tube cancer that did not respond to platinum chemotherapy (phase II closed as of 1/7/2011). Viral therapy may be able to kill tumor cells without damaging normal cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the safety and tolerability of intravenous (IV) and intraperitoneal (IP) administration of wild-type reovirus (REOLYSIN®).

II. Determine the maximum tolerated dose of IP REOLYSIN® when used with a fixed dose of IV REOLYSIN®.

III. Determine the objective response rate (complete response and partial response per Response Evaluation Criteria in Solid Tumors [RECIST] criteria) of treatment with IV and IP REOLYSIN® in patients with recurrent, platinum-refractory ovarian epithelial, peritoneal, or fallopian tube carcinoma. (Phase II) (phase II closed as of 1/7/2011).

SECONDARY OBJECTIVES:

I. To identify viral replication in tumor following IV reovirus. II. To identify anti-reovirus antibodies in patients being treated with IV and IP REOLYSIN® therapy.

III. To identify viral replication in the abdominal washings of patients undergoing IV and IP REOLYSIN® therapy.

IV. To correlate response to therapy with Ras oncogene status. V. To evaluate double-stranded RNA-activated protein kinase activity in tumors. VI. To correlate molecular predictors of response to REOLYSIN® therapy.

OUTLINE: This is a phase I, dose-escalation study of intraperitoneal (IP) wild-type reovirus when administered with fixed dose IV wild-type reovirus.

PHASE I: Patients receive wild-type reovirus IV over 60 minutes on days 1-5 in course 1, followed by insertion of an IP access port. Beginning in course 2, patients receive wild-type reovirus IV over 60 minutes on days 1-5 and wild-type reovirus IP over 10 minutes on days 1 and 2*. Treatment with IV and IP wild-type reovirus repeats every 28 days in the absence of disease progression or unacceptable toxicity.

PHASE II: Patients undergo IP access port insertion before beginning treatment. Patients receive wild-type reovirus IV over 60 minutes on days 1-5 and IP (at the maximum tolerated dose determined in phase I) over 10 minutes on days 1 and 2*. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity (phase II closed as of 1/7/2011). NOTE: *Patients receive IP wild-type reovirus on days 2 and 3 in course 3.

Prior to each IP wild-type reovirus administration, normal saline is administered through the IP catheter and withdrawn for correlative studies in courses 2 and 3 (phase I) or courses 1 and 2 (phase II). Patients also undergo a CT-guided percutaneous tumor biopsy on day 2 of course 3 (phase I or II). Samples are analyzed by immunohistochemistry, RT-PCR, and electron microscopy for the relevant molecular effects of wild-type reovirus on tumor and normal tissue.

After completion of study treatment, patients are followed for up to 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed ovarian epithelial, primary peritoneal, or fallopian tube cancer
* Recurrent disease after platinum-based chemotherapy

  * Must have experienced disease persistence during primary platinum-based therapy or recurrence within 12 months after completion of platinum-based chemotherapy ("platinum-refractory" or "platinum-resistant" disease)

    * A patient receiving a second course of platinum-based chemotherapy for platinum-sensitive disease who then develops persistence or recurrence within 12 months is considered eligible for this trial
* Must have measurable disease by RECIST criteria (phase II) (phase II closed as of 1/7/2011)
* Must have received ≥ 1 prior platinum-based cytotoxic chemotherapy regimen (for primary disease) containing carboplatin, cisplatin, or other organoplatinum compound

  * Initial treatment may have included any of the following:

    * High-dose therapy
    * Consolidation therapy
    * Intraperitoneal (IP) therapy
    * Extended therapy administered after surgical or nonsurgical assessment
  * One additional non-cytotoxic regimen (e.g., monoclonal antibodies, cytokines, or small-molecule inhibitors) for recurrent or persistent disease allowed
* Patients may have received hormonal therapy for management of disease (e.g., SERMs, aromatase inhibitors, progestins, and GnRH agonists)
* No loculated ascites for which IP distribution of virus is not expected to be feasible
* No known brain metastases
* GOG performance status (PS) 0-2 (Karnofsky PS 60-100%)
* Life expectancy > 12 weeks
* Leukocytes ≥ 3,000/mcL
* Absolute neutrophil count ≥ 1,500/mcL
* Hemoglobin ≥ 10 g/dL
* Platelets ≥ 100,000/mcL
* Total bilirubin normal
* AST/ALT ≤ 2.5 times upper limit of normal
* Creatinine normal
* Ejection fraction > 50% by echocardiogram or MUGA
* Cardiac enzymes normal
* Not pregnant or nursing
* Fertile patients must use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for the duration of study participation
* Must be able to avoid direct contact with pregnant or nursing women, infants, or immunocompromised individuals while on study and for ≥ 3 weeks following the last dose of study agent administration
* Cardiac conduction abnormalities (e.g., bundle branch block, heart block) are allowed if their cardiac status has been stable for 6 months before study entry
* At least 4 weeks since most recent cytotoxic chemotherapy (6 weeks for nitrosoureas or mitomycin C)
* Recovered from adverse events due to agents administered more than 4 weeks earlier
* No prior radiotherapy to the abdomen or pelvis
* No other concurrent investigational agents
* No investigational or commercial agents or therapies other than those described below may be administered with the intent to treat the patient's malignancy

Exclusion Criteria:

* Patients in whom insertion of an IP catheter is not feasible due to surgical contraindications or abdominal and pelvic adhesions
* Known HIV infection or hepatitis B or C
* Clinically significant cardiac disease (New York Heart Association class III or IV cardiac disease) including any of the following:

  * Pre-existing arrhythmia
  * Uncontrolled angina pectoris
  * Myocardial infarction 1 year prior to study entry
  * Compromised left ventricular ejection fraction ≥ grade 2 by MUGA or echocardiogram
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, or psychiatric illness/social situations that would limit compliance with study requirements
* Chronic oral steroids at an equivalent dose of prednisone 5 mg daily

  * Inhaled steroids allowed
* Patients on immunosuppressive therapy
* Concurrent routine prophylactic use of growth factor (filgrastim [G-CSF] or sargramostim [GM-CSF])

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2008-04; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Maximum tolerable dose of intraperitoneal (IP) wild-type reovirus when administered with fixed dose IV wild-type reovirus (phase I) | At each dose level, assessed up to 5 dose levels
  Dose-limiting toxicity will be assessed using the Common Terminology Criteria for Adverse Events (CTCAE) v. 4
Objective response (partial response and complete response) | Every 8 weeks during treatment and assessed up to 12 weeks after completion of treatment
  Response will be evaluated using the new international criteria proposed by RECIST Committee.

SECONDARY OUTCOMES:
Association of Ras oncogene and molecular markers with objective response | During courses 1 and 2, and prior to course 3
  Secondary endpoints are generally descriptive

CONTACTS AND LOCATIONS:
Overall Officials: David Cohn, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States